CLINICAL TRIAL: NCT06282848
Title: Pharmacological (0.05% Atropine) and Non-pharmacological (Defocused Incorporated Multiple Segments Lens) Treatment Effects on the Children With Different Predicted Myopia Progression Rate Measured by Modified Multifocal Electroretinogram
Brief Title: Pharmacological and Non-pharmacological Treatment Effects on Children With Different Predicted Myopia Progression Rate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry HL Chan, PhD, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HongKongPU_Optometry4
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Myopia; Atropine; Optical defocus; Electroretinogram; Retina
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine 0.05% (Active Comparator): Group receiving atropine treatment for 18 months after 6 months of monitoring without intervention
  Interventions: Drug: Atropine 0.05%
- DIMS lens (Experimental): Group receiving DIMS lens treatment for 18 months after 6 months of monitoring without intervention
  Interventions: Device: DIMS lens

INTERVENTIONS:
Drug: Atropine 0.05% — Topical application
  Arms: Atropine 0.05%
Device: DIMS lens — Spectacle wear
  Arms: DIMS lens

SUMMARY:
The goal of this clinical trial is to compare pharmacological and non-pharmacological treatment effects on the children with different predicted myopia progression rate measured by modified multifocal electroretinogram. The main questions it aims to answer are:

* the effectiveness of using 0.05% atropine and prescribing DIMS lens for myopia control in children with different myopia progression rates
* the contribution of L/M cones in juvenile myopia progression and changes of retinal activities under atropine and DIMS treatment.

Participants will have baseline and follow-up eye examinations and given either pharmacological treatment with 0.05% atropine or non-pharmacological treatment with DIMS lens for myopia control.

Researchers will compare the changes of refractive errors and axial length after different types of interventions and investigate the relations between the parameters of mfERG responses and the thicknesses of retinal layers and choroid.

DETAILED DESCRIPTION:
This proposed study is a 24-month longitudinal randomized trial that aims to investigate myopia development after either topical application of 0.05% atropine or prescription of DIMS lens in children with various predicted myopia progression rates by their initial retinal responses obtained by multifocal ERG. This will help elucidate the effectiveness of using 0.05% atropine and prescribing DIMS lens for myopia control in children with different myopia progression rates. The retinal electrophysiological investigation will help determine the contribution of L/M cones in juvenile myopia progression and changes of retinal activities under atropine and DIMS treatment.

80 subjects in either gender aged 7 to 9 years will be recruited in this study. They should have spherical equivalent refractive error between -0.5D and -4D in both eyes with best-corrected visual acuity of logMAR 0.00 or better. All should have normal eye health and without systemic diseases or epilepsy. They have not received any myopia control previously. Eligible subjects will have a baseline eye examination and have the first 6-month period monitoring the refractive and ocular changes compared with the baseline control data. After these 6 months, subjects will be classified into either fast or slow myopia progression group in accordance with the results of electrophysiology results and then will further be randomly allocated either intervention group: pharmacological treatment group (daily topical 0.05% atropine) or control group: non-pharmacological treatment group (daily wear of Defocused Incorporated Multiple Segments - DIMS lenses), for 18 months study period with 6-month interval regular follow up.

The primary outcomes are the changes of refractive errors and axial length after different types of interventions and the secondary outcomes are the relations between the parameters of mfERG responses and the thicknesses of retinal layers and choroid.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 7 and 9 years
* have no reported eye disorder and no family history of eye disease
* be able to participate in this study for 24 months
* not have any current or history of epilepsy
* not have any current or history of asthma
* have refractive error between 0.50 D and 4.00 D and less than 1.50D of astigmatism with best corrected visual acuity of LogMAR 0.0 or better
* have no detected eye diseases or disorders after eye examination, except myopia

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subjective refraction | up to 24 months
  Refractive error (in Diopter)
Axial length | up to 24 months
  Length of eyeball

SECONDARY OUTCOMES:
mfERG responses | up to 24 months
  Parameters of mfERG responses
Retinal and choroidal thickness | up to 24 months
  Thicknesses of retinal layers and choroid

CONTACTS AND LOCATIONS:
Overall Officials: Henry HL CHAN, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT06282848/ICF_000.pdf